CLINICAL TRIAL: NCT01204333
Title: Thrombolysis or Anticoagulation for Cerebral Venous Thrombosis (TOACT)
Brief Title: Thrombolysis or Anticoagulation for Cerebral Venous Thrombosis
Acronym: TOACT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jan Stam, MD, PhD (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Sponsor-Investigator, Jan Stam, MD, PhD, Prof. Dr. J. Stam, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOACT
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-11

CONDITIONS: Sinus Thrombosis, Intracranial
Keywords: Cerebral venous and sinus thrombosis; Cerebral venous thrombosis; Sinus Thrombosis, Intracranial; Endovascular thrombolysis; Thrombolysis; Thrombectomy
MeSH Terms: conditions — Sinus Thrombosis, Intracranial; Intracranial Thrombosis | interventions — Tissue Plasminogen Activator; Urokinase-Type Plasminogen Activator; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endovascular thrombolysis (Experimental)
  Interventions: Drug: Endovascular thrombolysis
- Standard treatment (Active Comparator)
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Endovascular thrombolysis — Endovascular thrombolysis consists of local application of alteplase or urokinase within the thrombosed sinuses. Standard endovascular techniques to mechanically remove clot material, such as thrombosuction, are allowed, but not mandatory.
  Other Names: Alteplase; Urokinase
  Arms: Endovascular thrombolysis
Drug: Heparin — The patients randomized to standard care will receive (or continue) either intravenous adjusted dose unfractionated heparin (aPTT value kept within 1.5 to 2.5 times the normal value), or any type of body-weight adjusted low molecular weight heparin in therapeutic dose, according to local custom and international guidelines
  Arms: Standard treatment

SUMMARY:
Background: Endovascular thrombolysis, with or without mechanical clot removal (ET), may be beneficial for a subgroup of patients with cerebral venous sinus thrombosis (CVT), who have a poor prognosis despite treatment with heparin. Published experience with ET is promising, but only based on case series and not on controlled trials.

Objective: The main objective of the TO-ACT trial is to determine if ET improves the functional outcome of patients with a severe form of CVT

Study design: The TO-ACT trial will be designed as a multi-centre, prospective, randomized, open-label, blinded endpoint (PROBE) trial.

Study population: Patients are eligible if they have a radiologically proven CVT, a high probability of poor outcome (defined by presence of one or more of the following risk factors: mental status disorder, coma, intracranial hemorrhagic lesion or thrombosis of the deep cerebral venous system) and the responsible physician is uncertain if ET or standard anti-coagulant treatment is better.

Intervention: Patients will be randomized to receive either ET or standard therapy (therapeutic doses of heparin). ET consists of local application of alteplase or urokinase within the thrombosed sinuses, and/or mechanical thrombectomy. Glasgow coma score, NIH stroke scale and relevant laboratory parameters will be assessed at baseline.

Endpoints: The primary endpoint is the modified Rankin scale (mRS) at 12 months. The most important secondary outcomes are the mRS, mortality and recanalization rate at 6 months. Major intra- and extracranial hemorrhagic complications within one week following the intervention are the principal safety outcome. Results will be analyzed according to the "intention-to-treat" principle. Assessment of study endpoints will be carried out according to standardized questionnaires by a blinded neurologist or research nurse who is not involved in the treatment of the patient.

Study size: To detect a 50% relative reduction in mRS≥2 (from 40 to 20%), 164 patients (82 in each treatment arm) have to be included (two-sided alpha, 80% power).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Included patients may benefit directly from ET. Complications of ET, most notably intracranial hemorrhages, constitute the most important risk of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Cerebral venous thrombosis, confirmed by cerebral angiography (with intra-arterial contrast injection), magnetic resonance venography or computed tomographic venography.
2. Severe form of CVT with a high chance of incomplete recovery, as defined by the presence of one or more of the following risk factors

   1. Intracerebral hemorrhagic lesion due to CVT
   2. Mental status disorder
   3. Coma (Glasgow coma scale < 9)
   4. Thrombosis of the deep cerebral venous system
3. Uncertainty by the treating physician if ET or standard heparin therapy is the optimal therapy for the patient.

Exclusion Criteria:

* Age less than 18 years
* Duration from diagnosis to randomization of more than 10 days
* Recurrent CVT
* Any thrombolytic therapy within last 7 days
* Pregnancy (women in the puerperium may be included)
* Isolated cavernous sinus thrombosis
* Isolated intracranial hypertension (without focal neurological signs, with the exception of papilloedema and 6th cranial nerve palsy)
* Cerebellar venous thrombosis with 4th ventricle compression and hydrocephalus, which requires surgery
* Contraindication for anti-coagulant or thrombolytic treatment

  1. documented generalized bleeding disorder
  2. concurrent thrombocytopenia (<100 x 10E9/L)
  3. documented severe hepatic or renal dysfunction, that interferes with normal coagulation
  4. uncontrolled severe hypertension (diastolic > 120 mm Hg)
  5. known recent (< 3 months) gastrointestinal tract hemorrhage (not including he¬morrhage from rectal hemorrhoids)
* Any known associated condition (such as terminal cancer) with a poor short term (1 year) prognosis independent of CVT
* Clinical and radiological signs of impending transtentorial herniation due to large space-occupying lesions (e.g. large cerebral venous infarcts or hemorrhages)
* Recent (< 2 weeks) major surgical procedure (does not include lumbar puncture) or severe cranial trauma
* Known allergy against contrast fluid used during endovascular procedures or the thrombolytic drug used in that particular centre
* Previously legally incompetent prior to CVT
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-09; Primary Completion 2016-12 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Favorable clinical outcome (modified Rankin score 0-1) | 12 months after randomization
  Outcome on the modified Rankin Scale (mortality included) at 12 months after randomization is considered the primary study outcome to determine the efficacy of thrombolytic treatment. For the primary endpoint the mRS will be dichotomized between 1 and 2 (i.e. incomplete recovery is defined as a score of 2 or higher, including death).

SECONDARY OUTCOMES:
Favorable clinical outcome (modified Rankin score 0-1) | 6 months after randomization
Recanalization rate of cerebral venous system | 6 months
All cause mortality | 6 months
Required surgical intervention in relation to CVT | 6 months
  The proportion of surgical intervention that are required in relation to cerebral venous thrombosis (e.g. ventricular shunting procedures or craniotomy)
Major extracranial and symptomatic intracranial hemorrhagic complications | 1 week after randomization
  Extracranial hemorrhage is classified as major if clinically overt and associated with fall in hemoglobin of 1.2 mmol/l (2 gram/dl) or more within 48 hours, if it is retroperitoneal, intracranial or intraocular, or requires a transfusion of two or more units of packed cells. Any bleeding requiring operation or leading to death is regarded as major. Symptomatic intracranial hemorrhage is defined as any apparently extravascular blood in the brain associated with an increase of 4 points or more on the NIHSS score, or leading to death.
Dead or dependency (modified Rankin score 3-6) | 6 and 12 months
Modified Rankin Scale at 1 month after randomization | 1 month after randomization

OTHER OUTCOMES:
Interim analyses: Favorable clinical outcome (modified Rankin score 0-1) | After inclusion of 1/3rd and 2/3rd of patients
  The DSMB will perform two interim analyses after 55 and 110 patients (1/3rd and 2/3rd of all patients) have been randomized and completed the 12-month follow-up evaluation. As a stopping rule for efficacy, the Haybittle-Peto method will be used:
  * Interim analysis 1: p = 0,001
  * Interim analysis 2: p = 0,001
  In addition, the DSMB will assess futility during the interim analyses. The trial will be discontinued for futility if the conditional power (or probability of observing a statistically significant result in favor of the intervention group given the data obtained so far) is below 20%. This conditional power will be calculated under the assumption that in the remaining two-thirds/one-thirds of the study population the distributions of the primary endpoint will be the same as observed at the interim analysis.
  For the interim analyses the DSMB will use the primary outcome measure (modified Rankin score 0-1 at 12 months) for the determination of efficacy and futility.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stam, MD, PhD, Study Chair — University of Amsterdam; Jose M Ferro, MD, PhD, Principal Investigator — Hospital Santa Maria, Lisbon, Portugal; Marie-Germaine Bousser, MD, PhD, Principal Investigator — Hôpital Lariboisière, Paris, France; Patricia Canhão, MD, PhD, Principal Investigator — Hospital Santa Maria, Lisbon, Portugal; Isabelle Crassard, MD, PhD, Principal Investigator — Hôpital Lariboisière, Paris, France; Charles BL Majoie, MD, PhD, Principal Investigator — University of Amsterdam; Jim A Reekers, MD, PhD, Principal Investigator — University of Amsterdam; E Houdart, MD, PhD, Principal Investigator — Hôpital Lariboisière, Paris, France; Rob J de Haan, PhD, Principal Investigator — University of Amsterdam
Locations (15):
- Centre hospitalier de l'université de Montréal (CHUM), Montreal, Canada
- XuanWu Hospital, Beijing, China
- Hôpital Lariboisière, Paris, France
- Netherlands (6):
  - Academic Medical Centre, Amsterdam
  - University Medical Centre Groningen, Groningen
  - St. Antonius hospital, Nieuwegein
  - Erasmus Medical Centre, Rotterdam
  - Haga hospital, The Hague
  - Medical Centre Haaglanden, The Hague
- Portugal (5):
  - Hospital de Braga, Braga
  - Hospital da Universidade de Coimbra, Coimbra
  - Hospital Santa Maria, Lisbon
  - Hospital Sao Jose hospital, Lisbon
  - Hospital de Santo António, Porto
- Inselspital, University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Coutinho JM, Stam J. How to treat cerebral venous and sinus thrombosis. J Thromb Haemost. 2010 May;8(5):877-83. doi: 10.1111/j.1538-7836.2010.03799.x. Epub 2010 Feb 9. PMID 20149074
- [Background] Canhao P, Falcao F, Ferro JM. Thrombolytics for cerebral sinus thrombosis: a systematic review. Cerebrovasc Dis. 2003;15(3):159-66. doi: 10.1159/000068833. PMID 12646773
- [Background] Ciccone A, Canhao P, Falcao F, Ferro JM, Sterzi R. Thrombolysis for cerebral vein and dural sinus thrombosis. Cochrane Database Syst Rev. 2004;2004(1):CD003693. doi: 10.1002/14651858.CD003693.pub2. PMID 14974030
- [Background] Stam J, Majoie CB, van Delden OM, van Lienden KP, Reekers JA. Endovascular thrombectomy and thrombolysis for severe cerebral sinus thrombosis: a prospective study. Stroke. 2008 May;39(5):1487-90. doi: 10.1161/STROKEAHA.107.502658. Epub 2008 Mar 13. PMID 18340091
- [Derived] Coutinho JM, Zuurbier SM, Bousser MG, Ji X, Canhao P, Roos YB, Crassard I, Nunes AP, Uyttenboogaart M, Chen J, Emmer BJ, Roosendaal SD, Houdart E, Reekers JA, van den Berg R, de Haan RJ, Majoie CB, Ferro JM, Stam J; TO-ACT investigators. Effect of Endovascular Treatment With Medical Management vs Standard Care on Severe Cerebral Venous Thrombosis: The TO-ACT Randomized Clinical Trial. JAMA Neurol. 2020 Aug 1;77(8):966-973. doi: 10.1001/jamaneurol.2020.1022. PMID 32421159
- [Derived] Coutinho JM, Ferro JM, Zuurbier SM, Mink MS, Canhao P, Crassard I, Majoie CB, Reekers JA, Houdart E, de Haan RJ, Bousser MG, Stam J. Thrombolysis or anticoagulation for cerebral venous thrombosis: rationale and design of the TO-ACT trial. Int J Stroke. 2013 Feb;8(2):135-40. doi: 10.1111/j.1747-4949.2011.00753.x. Epub 2012 Feb 20. PMID 22340437